CLINICAL TRIAL: NCT06946966
Title: The Effects of Online Mat Pilates and Face-to-Face Equipment-Based Pilates on Pain, Kinesiophobia, and Balance in Individuals With Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-04/02
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain
Keywords: pain
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reformer Pilates (Experimental): Reformer Pilates
  Interventions: Other: Reformer Pilates
- Pilates control (Active Comparator): Pilates control
  Interventions: Other: Pilates control
- pilates online pilates (Active Comparator): online pilates
  Interventions: Other: pilates online pilates

INTERVENTIONS:
Other: Reformer Pilates — Reformer Pilates
  Arms: Reformer Pilates
Other: Pilates control — Pilates control
  Arms: Pilates control
Other: pilates online pilates — pilates online pilates
  Arms: pilates online pilates

SUMMARY:
Non-specific low back pain (NSLBP) is a common musculoskeletal condition that affects a significant portion of the population and often leads to limitations in daily activities, reduced quality of life, and increased levels of kinesiophobi

DETAILED DESCRIPTION:
compare the effects of online mat Pilates and face-to-face equipment-based Pilates on pain, kinesiophobia, and balance in individuals with NSLBP. While both methods emphasize neuromuscular control and alignment, differences in delivery modes and equipment usage may influence outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years
* Non-specific low back pain for more than 12 weeks
* No clear pathological diagnosis
* Physically and cognitively capable of performing the exercises
* Pain level between 3 and 7 on the Visual Analog Scale (VAS)

Exclusion Criteria:

* Pregnancy
* Spinal surgery in the last 6 months
* Neurological or chronic systemic diseases
* Movement restriction due to severe pain

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
visual pain scal | 12 weeks
  A 10-cm line where participants mark their pain intensity, ranging from 'no pain' to 'worst pain'.
Quebec Back Pain Disability Scale (QBPDS) | 12 weeks
  Assesses functional disability related to back pain through 20 daily activity items. Higher scores indicate greater limitation in performing physical tasks.
Pressure Algometer | 12 weeks
  Measures the minimum pressure that causes pain in a specific muscle or soft tissue, helping to quantify pain sensitivity objectively.
Y-Balance Test (YBT) | 12 weeks
  Evaluates balance by measuring reach distance in three directions while standing on one leg. It reflects dynamic stability, core control, and lower limb function.
Tampa Scale of Kinesiophobia (TSK) | 12 weeks
  Assesses fear of movement and re-injury through a 17-item questionnaire. Higher scores indicate increased avoidance behavior and movement-related fear.The final score can be a minimum of 17 points and a maximum of 68 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahceşehir University Health Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No